CLINICAL TRIAL: NCT02107274
Title: Efficacy of Azithromycin in Treatment of Bronchiectasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, ALBERT IRUTHIARAJ L. ANTHONY, DR, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMRR-09-1075-5016
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Bronchiectasis
Keywords: Azithromycin; Bronchiectasis; Macrolide; Inflammation; Pulmonary
MeSH Terms: conditions — Bronchiectasis; Inflammation | interventions — Azithromycin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin and Placebo for Azithromycin (Active Comparator): Patients randomised to the treatment arm are to receive 1000 mg of azithromycin once a week for 12 weeks followed by placebo for azithromycin once weekly for another 12 weeks
  Interventions: Drug: Azithromycin
- Placebo for Azithromycin (Placebo Comparator): In Part One of the study participants will be randomised to receive 12 weeks of either placebo or azithromycin in a 1:1 ratio in a double-blinded fashion. After 12 weeks, in Part Two of the study, all participants will receive placebo in a double-blinded fashion for an additional 12 weeks.
  Interventions: Drug: Placebo for Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin (C38H72N2O12 MW 749) is a 15-membered azalide, a subclass of macrolide antibiotics
  Other Names: Zithromax 250 mg tablet
  Arms: Azithromycin and Placebo for Azithromycin
Drug: Placebo for Azithromycin — In Part One of the study participants will be randomised to receive 12 weeks of either placebo or azithromycin in a 1:1 ratio in a double-blinded fashion. After 12 weeks, in Part Two of the study, all participants will receive placebo in a double-blinded fashion for an additional 12 weeks.
  Arms: Placebo for Azithromycin

SUMMARY:
Bronchiectasis is a chronic lung condition characterised primarily by dilatation of the airways. Only a small number of clinical studies have been conducted investigating the use of macrolides to treat non-cystic fibrosis bronchiectasis. The purpose of this study is to determine the efficacy of 12 weeks treatment with azithromycin in adult patients with non-cystic fibrosis bronchiectasis.

DETAILED DESCRIPTION:
Previous studies of various macrolides with small sample sizes have reported some benefit with the reduction of sputum volume in bronchiectasis patients. However, macrolide therapy could not yet be confidently used to treat bronchiectasis, given the diffuse nature of these findings. These studies have had a wide range of hypotheses, and have not necessarily focused on the anti-inflammatory effects of macrolides. Furthermore, these studies are few in number, and not all have been placebo-controlled or double-blinded. This, combined with the small sample sizes used, limits the reliability of these results. This study aims to expand on these limited published findings by investigating a larger sample population with different endpoints. Sputum volume and quality of life have been selected as important variables to aid in assessing efficacy.

This study aims to be independent of previous studies in a number of ways. This is the only study of bronchiectasis patients to formally investigate quality of life after treatment with a macrolide, and the potential carryover effect of azithromycin therapy. This study will also expand on the findings of previous studies of macrolides in bronchiectasis by incorporating a larger sample size into the trial.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent to participate in the study in accordance with the local ethics committee regulations
* Have a confirmed diagnosis of bronchiectasis (by HRCT) Aged 18 years or over Have chronic sputum production, defined as a greater than 45 mililitres volume produced in the 1 week prior to study entry.
* Be able to perform reproducible spirometry
* Be in a relatively stable disease state in the 6 weeks prior to entry, as defined by the absence of the following: respiratory exacerbations requiring hospitalisation, change in cough and/or sputum production, new or increased hemoptysis, more than 10% weight loss, use of additional antibiotic courses

Exclusion Criteria:

* Subjects will be excluded if one or more of the following criteria occur. The subject: Is an investigator, or an immediate family member of an investigator
* Has a confirmed diagnosis of cystic fibrosis, as evidenced by genetic analysis or a sweat test result more than 60mmol/L
* Has a primary immunodeficiency Is a pregnant or lactating female Has had a respiratory exacerbation requiring hospitalisation or additional course of antibiotics in the 6 weeks prior to study entry
* Has been prescribed or used oral steroids on any occasion for the 3 months prior to study entry.
* Has been using mucolytic agents on any occasion for the 2 months prior to study entry Has active tuberculosis
* Has an active malignancy, including melanoma (other skin carcinomas excluded)
* Has a history of significant liver disease or insufficiency Has a significant history of drug abuse (including alcohol abuse) or mental illness Has a known intolerance or allergy to macrolides
* Has been participating in another interventional drug study in the 3 months prior to enrolment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALBERT IRUTHIARAJ ANTHONY, MBBS, Principal Investigator — Penang Hospital, Malaysia
Locations (1):
- Respiratory Unit, Taiping Hospital, Taiping, Perak, Malaysia

REFERENCES:
- [Background] Cymbala AA, Edmonds LC, Bauer MA, Jederlinic PJ, May JJ, Victory JM, Amsden GW. The disease-modifying effects of twice-weekly oral azithromycin in patients with bronchiectasis. Treat Respir Med. 2005;4(2):117-22. doi: 10.2165/00151829-200504020-00005. PMID 15813663
- [Background] Anwar GA, Bourke SC, Afolabi G, Middleton P, Ward C, Rutherford RM. Effects of long-term low-dose azithromycin in patients with non-CF bronchiectasis. Respir Med. 2008 Oct;102(10):1494-6. doi: 10.1016/j.rmed.2008.06.005. Epub 2008 Jul 23. PMID 18653323
- [Background] Davies G, Wilson R. Prophylactic antibiotic treatment of bronchiectasis with azithromycin. Thorax. 2004 Jun;59(6):540-1. No abstract available. PMID 15170047
- [Derived] Lourdesamy Anthony AI, Muthukumaru U. Efficacy of azithromycin in the treatment of bronchiectasis. Respirology. 2014 Nov;19(8):1178-82. doi: 10.1111/resp.12375. Epub 2014 Sep 2. PMID 25183304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 subjects with a High Resolution CT scan diagnosis of pulmonary bronchiectasis was recruited from January - October 2011. Recruitment was done amongst patients in chest clinic, Hospital Taiping. A total of 78 subjects were selected based on the inclusion and exclusion criterias.
Pre-assignment Details: 12 subjects were excluded from randomization as they did not have chronic sputum production and were unable to perform spirometry.
Groups:
- Azithromycin and Placebo for Azithromycin: Patients randomised to the treatment arm received 1000mg of azithromycin once a week for 12 weeks followed by placebo for azithromycin once a week for another 12 weeks.
- Placebo for Azithromycin: Patients randomised to the control arm received placebo for azithromycin once a week for 12 weeks followed by placebo for azithromycin once a week for another 12 weeks.
Period: Treatment vs. Placebo
Arm/Group | Azithromycin and Placebo for Azithromycin | Placebo for Azithromycin
Started | 39 | 39
Completed | 36 | 37
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 2
Period: Control Phase
Arm/Group | Azithromycin and Placebo for Azithromycin | Placebo for Azithromycin
Started | 36 | 37
Completed | 33 | 35
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 2 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Azithromycin: Patients randomised to the treatment arm received 1000mg of azithromycin once a week for 12 weeks followed by placebo for azithromycin once a week for another 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo for Azithromycin | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (11.77) | 59.7 (15.03) | 62.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 15 | 13 | 28
Sputum volume [Mean (Standard Deviation); unit: gram] — Higher sputum volume indicates active disease process and poorer morbidity. Lower sputum volume is associated with better control of disease process.
  gram | 41.8 (26.05) | 23.6 (20.67) | 32.4 (24.99)
St George's Respiratory Questionnaire (SGRQ) score [Mean (Standard Deviation); unit: Scores on a scale] — St George's Respiratory Questionnaire (SGRQ) score measures quality of life in patients with chronic lung disease. Score can range from 10 (minimum) until 100 (maximum). Lower scores are associated with good quality of life and the higher scores indicates poor quality of life. Total score is a product of summation of individual scores per question.
  Scores on a scale | 41.06 (9.95) | 36.40 (10.59) | 38.66 (10.47)
Forced Expiratory Volume at 1 second (FEV1) [Mean (Standard Deviation); unit: Litres] — Forced expiratory volume at 1 second (FEV1) is a reflection of lung volume. Higher values reflect less airflow limitation and good lung reserve. Lower values indicate poor airflow limitation and lower lung reserve.
  Litres | 1.08 (0.41) | 1.17 (0.54) | 1.13 (0.48)
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: Litres] — Forced vital capacity (FVC) is a measurement of lung volume. Higher values reflect better reserve meanwhile lower values indicate poorer reserve.
  Litres | 1.56 (0.65) | 1.69 (0.74) | 1.63 (0.70)

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Sputum Volume
Description: Each participant must be instructed and enabled to collect 24 hour sputum volumes over the 24 hours prior to visits 3, 6 and 8, inclusive. As this is the primary endpoint of the study, it is critical that 24 hour sputum volumes are measured and recorded accurately, observing the following protocol: The subject should be given a sterile jar to collect the sputum, which has been weighed previously for convenience. Each jar will be labelled with subject name, start and finish time/date The collection should commence on rising in the morning and complete 24 hours later. Ensure that the sputum sample has minimal saliva in the collection Instruct subject to collect all sputum produced spontaneously or after coughing over a single daytime 24 hour period. The sample should come from the lungs and should not be salivary. Encourage subject not to swallow sputum, but to collect. Each 24 hour collection period should be as similar as possible in terms of physiotherapy and exercise regimens
Time Frame: Visit 3 (Baseline); Visit 6 (Week 12); Visit 8 (Week 24)
Population: A total of 90 subjects were recruited. Among them, 78 subjects fulfilled the inclusion criteria and were randomized. Only 68 subjects completed the study and were subjected for analysis. We targeted to recruit 80 subjects and a dropout rate of 20% was anticipated as stated in the protocol.
Measure: Mean (Standard Deviation); unit: gram
Groups:
- Azithromycin: Patients randomised to the treatment arm received1000mg of azithromycin once a week for 12 weeks followed by placebo for azithromycin once a week for another 12 weeks.
Arm/Group | Azithromycin | Placebo for Azithromycin
Number analyzed (Participants) | 33 | 35
gram
  Visit 3(Baseline) | 41.8 (26.1) | 23.6 (20.7)
  Visit 6(Week 12) | 29.9 (19.4) | 26.2 (20.5)
  Visit 8(Week 24) | 30.4 (20.6) | 28.5 (21.6)
Statistical Analysis 1: Comparison: Azithromycin; Sputum volume were compared between Visit 6 (Week 12) and Visit 3 (Baseline), Visit 8 (Week 24) and Visit 3 (Baseline), as well for Visit 8 (Week 24) and Visit 6 (Week 12). Independent t-test was applied for study end points which were numerical variables; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — P value of less than 0.05 was considered as significant
Statistical Analysis 2: Comparison: Placebo for Azithromycin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — P value of less than 0.05 was considered significant

2. Secondary Outcome: Health Status: St George's Respiratory Questionnaire Score
Description: The St. George Respiratory Questionnaire is to be administered at visits 3, 6 and 8 inclusive. It should be administered in a quiet room where the participant can answer the questions without interruption, prior to any other protocol related procedures
Time Frame: Visit 3 (Baseline); Visit 6 (Week 12); Visit 8 (Week 24)
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Azithromycin | Placebo for Azithromycin
Number analyzed (Participants) | 33 | 35
Units
  Visit 3(Baseline) | 41.1 (9.9) | 36.4 (10.6)
  Visit 6(Week 12) | 30.2 (8.5) | 39.1 (9.3)
  Visit 8(Week 24) | 31.7 (8.1) | 41.1 (11.1)
Statistical Analysis 1: Comparison: Azithromycin; SGRQ scores were compared between Visit 6 (Week 12) and Visit 3 (Baseline), Visit 8 (Week 24) and Visit 3 (Baseline), as well for Visit 8 (Week 24) and Visit 6 (Week 12). Independent t-test was applied for study end points which were numerical variables; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — P value of less than 0.05 was considered as significant
Statistical Analysis 2: Comparison: Placebo for Azithromycin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — p valu of less than 0.05 was considered significant

3. Secondary Outcome: Spirometry Value; Forced Expiratory Volume at 1 Second (FEV1)
Description: Pulmonary function testing using a spirometer will be carried out at visits 3, 6 and 8 inclusive. All testing should be done in the sitting position, except for obese patients, who commonly obtain deeper inspiration when tested in the standing position. Subjects should avoid the following prior to lung function testing: Smoking within 1 hour of testing Consuming alcohol within 4 hours of testing Performing vigorous exercise within 30 minutes of testing Wearing restrictive clothing around the chest or abdomen Eating a large meal within 2 hours of testing The following medications must be withheld prior to testing, with the minimum time from last dose indicated- short acting beta agonists (6 hours), long acting beta agonists (12 hours), ipratropium bromide (12 hours), antihistamines (12 hours), long acting bronchodilator combinations (12 hours)
Time Frame: Visit 3 (Baseline); Visit 6 (Week 12); Visit 8 (Week 24)
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Azithromycin | Placebo for Azithromycin
Number analyzed (Participants) | 33 | 35
Litres
  Visit 3(Baseline) | 1.08 (0.41) | 1.17 (0.55)
  Visit 6(Week 12) | 1.09 (0.40) | 1.10 (0.53)
  Visit 8(Week 24) | 1.04 (0.37) | 1.08 (0.49)
Statistical Analysis 1: Comparison: Azithromycin; FEV1 values were compared between Visit 6 (Week 12) and Visit 3 (Baseline), Visit 8 (Week 24) and Visit 3 (Baseline), as well for Visit 8 (Week 24) and Visit 6 (Week 12). Independent t-test was applied for study end points which were numerical variables; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — P value of less than 0.05 was considered as significant
Statistical Analysis 2: Comparison: Placebo for Azithromycin; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — p value of less than 0.05 was considered significant

4. Secondary Outcome: Spirometric Values: Forced Vital Capacity (FVC)
Description: Pulmonary function testing using a spirometer will be carried out at visits 3, 6 and 8 inclusive. All testing should be done in the sitting position, except for obese patients, who commonly obtain deeper inspiration when tested in the standing position. Subjects should avoid the following prior to lung function testing: Smoking within 1 hour of testing Consuming alcohol within 4 hours of testing Performing vigorous exercise within 30 minutes of testing Wearing restrictive clothing around the chest or abdomen Eating a large meal within 2 hours of testing The following medications must be withheld prior to testing, with the minimum time from last dose indicated- short acting beta agonists (6 hours), long acting beta agonists (12 hours), ipratropium bromide (12 hours), antihistamines (12 hours), Iong acting bronchodilator combinations (12 hours)
Time Frame: Visit 3 (Baseline); Visit 6 (Week 12); Visit 8 (Week 24)
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Azithromycin | Placebo for Azithromycin
Number analyzed (Participants) | 33 | 35
Litres
  Visit 3(Baseline) | 1.56 (0.65) | 1.69 (0.74)
  Visit 6(Week 12) | 1.58 (0.63) | 1.60 (0.70)
  Visit 8(Week 24) | 1.55 (0.66) | 1.58 (0.72)
Statistical Analysis 1: Comparison: Azithromycin; FVC values were compared between Visit 6 (Week 12) and Visit 3 (Baseline), Visit 8 (Week 24) and Visit 3 (Baseline), as well for Visit 8 (Week 24) and Visit 6 (Week 12). Independent t-test was applied for study end points which were numerical variables; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — P value of less than 0.05 was considered as significant
Statistical Analysis 2: Comparison: Placebo for Azithromycin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — p value of less than 0.05 was considered significant

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse drug reactions for 24 weeks. Monitoring included enquiry of symptoms, physical examination and venous sampling at every visit.
Description: Any clinically significant result outside normal ranges from these visits was documented and was reported as an adverse event. The subjects were withdrawn from the trial and then monitoring will continue until resolution or an appropriate medical judgment has been made to determine the cause and severity of the case.
Arm/Group | Azithromycin | Placebo for Azithromycin
Serious Adverse Events (participants affected / at risk) | 5/33 | 4/35
Other Adverse Events (participants affected / at risk) | 3/33 | 1/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=33) | Placebo for Azithromycin (N=35)
Pneumonia Hospitalisations (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pneumonia Deaths (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=33) | Placebo for Azithromycin (N=35)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) — The diarrhea resolved upon discontinuation of study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes